CLINICAL TRIAL: NCT00717288
Title: Transitioning Post-cardiothoracic Surgery Patients From Intravenous Insulin to the Subcutaneous Route With Insulin Detemir.
Brief Title: Transitioning Open Heart Surgery Patients From Insulin Infusions to Detemir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Kathleen Dungan, Assistant Professor of Medicine, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007H0210; 60016576 (Other: Other)
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; hyperglycemia; open heart surgery; cardiothoracic surgery; detemir; insulin infusion; intravenous insulin
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia | interventions — Insulin Detemir

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Detemir insulin dosed at 50% of calculated basal insulin infusion requirement injected once daily
  Interventions: Drug: Detemir
- 2 (Active Comparator): Detemir insulin dosed at 65% of calculated basal insulin infusion requirement injected once daily
  Interventions: Drug: Detemir
- 3 (Active Comparator): Detemir insulin dosed at 80% of calculated basal insulin infusion requirement injected once daily
  Interventions: Drug: Detemir

INTERVENTIONS:
Drug: Detemir — Detemir dosed at 50% of calculated basal insulin infusion requirements
  Other Names: Levemir
  Arms: 1
Drug: Detemir — Detemir dosed at 65% of calculated basal insulin infusion requirements
  Arms: 2
Drug: Detemir — Detemir dosed at 80% of calculated basal insulin infusion requirements
  Arms: 3

SUMMARY:
In this study we will determine the proper method for transitioning patients from a continuous insulin infusion to periodic injections of a newer long-acting insulin called detemir (Levemir).

DETAILED DESCRIPTION:
High sugar (glucose) is common after surgery, even in patients who do not have diabetes. High glucose contributes to severe hospital complications and even death. Insulin infusions appear to reduce this risk, but are generally only continued for a few days after surgery. In this study, we will determine the proper method for transitioning patients from a continuous insulin infusion to periodic injections of a newer long-acting insulin called detemir (Levemir). 90 patients who have undergone recent open heart surgery and are requiring an insulin infusion will be enrolled. They will be randomly assigned to one of three doses of detemir, which consists of 50%, 65%, or 80% of the total daily insulin infusion requirement in the fasting state. Subjects will also receive identical mealtime coverage according to the amount of carbohydrate (glucose) that is ingested. It is expected that the high dose group will achieve superior glycemic control without excessive hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus
* post-cardiothoracic surgery
* requiring an insulin infusion of at least 1 unit/hour
* Age 18-75

Exclusion Criteria:

* Glucocorticoids
* total parenteral nutrition (TPN) or tube feeds
* Pregnancy
* Surgical procedures in the next 48 hours for whom intravenous (IV) insulin will be expected
* Expected length of stay less than 48 hours following cessation of the insulin drip
* Patients using subcutaneous insulin pumps
* Diabetic ketoacidosis
* End-stage renal disease
* End-stage liver disease
* Coma
* Potentially sensitive admissions: prisoners, human immunodeficiency virus(HIV), suicidality
* Unable to give consent in English

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-07; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Dungan, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 50% Conversion Factor: Detemir insulin dosed at 50% of calculated basal insulin infusion requirement injected once daily
- 65% Conversion Factor: Detemir insulin dosed at 65% of calculated basal insulin infusion requirement injected once daily
- 80% Conversion Factor: Detemir insulin dosed at 80% of calculated basal insulin infusion requirement injected once daily
Period: Overall Study
Arm/Group | 50% Conversion Factor | 65% Conversion Factor | 80% Conversion Factor
Started | 28 | 29 | 25
Completed | 28 | 29 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 50% Conversion Factor | 65% Conversion Factor | 80% Conversion Factor | Total
Number analyzed (Participants) | 28 | 29 | 25 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 24 | 19 | 65
  >=65 years | 6 | 5 | 6 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 58 (8.0) | 57 (9.1) | 61 (7.6) | 58.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 8 | 17
  Male | 23 | 25 | 17 | 65
Region of Enrollment [Number; unit: participants]
  United States | 28 | 29 | 25 | 82

OUTCOME MEASURES:

1. Primary Outcome: Patients With Morning (AM) Glucose Between 80-130 mg/dl on Day 2 and 3
Description: Number of patients with a morning glucose between 80-130 mg/dl on day 2 and day 3
Time Frame: day 2, day 3
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | 50% Conversion Factor | 65% Conversion Factor | 80% Conversion Factor
Number analyzed (Participants) | 28 | 29 | 25
participants | 10 | 18 | 14

2. Secondary Outcome: Patients With Hypoglycemia (Defined as Glucose <65 mg/dl)
Description: Number of patients with hypoglycemia (defined as glucose <65 mg/dl)
Time Frame: 48 hours
Population: Intention to treat (ITT)
Measure: Number; unit: participants
Groups:
- 50% Conversion Factor; 65% Conversion Factor; 80% Conversion Factor: Number of subjects with a BG value <65 mg/dl
Arm/Group | 50% Conversion Factor | 65% Conversion Factor | 80% Conversion Factor
Number analyzed (Participants) | 28 | 29 | 25
participants | 0 | 6 | 3

3. Secondary Outcome: Reversion to Intravenous Insulin for Failure of Glycemic Control
Description: Number of participants who went back on intravenous insulin for failure of glycemic control.
Time Frame: 72 hours
Measure: Number; unit: participants
Groups:
- 50% Conversion Factor; 65% Conversion Factor; 80% Conversion Factor: Number of subjects that reverted back to an insulin drip
Arm/Group | 50% Conversion Factor | 65% Conversion Factor | 80% Conversion Factor
Number analyzed (Participants) | 28 | 29 | 25
participants | 2 | 0 | 1

ADVERSE EVENTS:
Arm/Group | 50% Conversion Factor | 65% Conversion Factor | 80% Conversion Factor
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29 | 1/25
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 50% Conversion Factor (N=28) | 65% Conversion Factor (N=29) | 80% Conversion Factor (N=25)
Death (General disorders) | 0 (0) | 0/28 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50% Conversion Factor (N=28) | 65% Conversion Factor (N=29) | 80% Conversion Factor (N=25)
BG <40 mg/dl (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) — Any BG <40 mg/dl

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No